CLINICAL TRIAL: NCT05482841
Title: Lung Ultrasound Score After Ear, Nose and Throat Cancer Surgery
Brief Title: Lung Ultrasound Score After ENT Cancer Surgery
Acronym: LUSENT
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: LUSENT
Record Dates: First submitted 2022-06-23; First posted 2022-08-01 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cancer of Head and Neck; Tracheostomy; Postoperative Pulmonary Complication; Surgery
Keywords: Postoperative pulmonary complication; Lung ultrasound; Tracheostomy; ENT cancer surgery
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ENT cancer surgery patients: all patients undergoing ENT cancer surgery with tracheotomy or tracheostomy at the Centre Léon Bérard.
  Interventions: Diagnostic Test: Lung ultrasound score

INTERVENTIONS:
Diagnostic Test: Lung ultrasound score — To evaluate the incidence of pulmonary atelectasis in the post-anesthesia care unit (PACU) using lung ultrasound.

SUMMARY:
After ENT cancer surgery, postoperative respiratory complications are common, especially after tracheostomy.

The objective of this study is to characterize the pulmonary status of patients after ENT cancer surgery.

We wish to collect and analyze the pulmonary abnormalities revealed by the ultrasound scans performed in the post-anesthesia care unit (PACU), at day 1 and at day 2 after ENT cancer surgery with tracheostomy.

DETAILED DESCRIPTION:
After ENT cancer surgery, postoperative respiratory complications are common, especially after tracheostomy.

Problems with lung ventilation called "atelectasis" are largely associated with these complications. These atelectasis develop within minutes of the start of general anesthesia. Patients who develop a complication require longer postoperative oxygen treatment and more physical therapy.

The diagnosis of atelectasis can be made by standard chest radiography, which is a source of radiation and requires moving the patient. An alternative technique, lung ultrasound, is a non-irradiating examination that can be performed in the patient's bed. It is routinely performed in the postoperative surveillance room and in the intermediate care unit at the Centre Léon Bérard.

The objective of this study is to characterize the pulmonary status of patients after ENT cancer surgery.

We wish to collect and analyze the pulmonary abnormalities revealed by the ultrasound scans performed in the post-anesthesia care unit (PACU), at day 1 and at day 2 after ENT cancer surgery with tracheostomy.

ELIGIBILITY:
Inclusion Criteria:

* ENT cancer surgery with tracheostomy or tracheotomy

Exclusion Criteria:

* under 18 years old
* deprivation of liberty
* pre-existing tracheotomy or tracheostomy
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ENT cancer surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasound score, in the PACU after ENT cancer surgery. | Up to 24 hours
  Lung ultrasound score : Images were obtained in PACU. Care was taken to set the focal zone on the pleural line. The thorax was divided into 12 quadrants: anterior, lateral, and posterior zones (separated by the anterior and posterior axillary lines) each divided in upper and lower portions for the right and left lung. Intercostal spaces of each of these areas were scanned and a cine-loop of the most pathologic area of each quadrant was saved to digital format.
  A semiquantitative score, the lung ultrasound (LUS) score, was calculated to assess lung aeration at each time point as described by Monastesse.

SECONDARY OUTCOMES:
Lung ultrasound score, on day 2 after ENT cancer surgery. | on the 2nd day after surgery
  Lung ultrasound score : Images were obtained on day 2 after PACU (in intermediate care unit). Care was taken to set the focal zone on the pleural line. The thorax was divided into 12 quadrants: anterior, lateral, and posterior zones (separated by the anterior and posterior axillary lines) each divided in upper and lower portions for the right and left lung. Intercostal spaces of each of these areas were scanned and a cine-loop of the most pathologic area of each quadrant was saved to digital format.
  A semiquantitative score, the lung ultrasound (LUS) score, was calculated to assess lung aeration at each time point as described by Monastesse.
Lung ultrasound score, on day 1 after ENT cancer surgery. | on the 1st day after surgery
  Lung ultrasound score : Images were obtained on day 1 after PACU (in intermediate care unit). Care was taken to set the focal zone on the pleural line. The thorax was divided into 12 quadrants: anterior, lateral, and posterior zones (separated by the anterior and posterior axillary lines) each divided in upper and lower portions for the right and left lung. Intercostal spaces of each of these areas were scanned and a cine-loop of the most pathologic area of each quadrant was saved to digital format.
  A semiquantitative score, the lung ultrasound (LUS) score, was calculated to assess lung aeration at each time point as described by Monastesse.
To assess the incidence of pulmonary atelectasis in the PACU by chest radiography. | Up to 24 hours
  pulmonary atelectasis on chest radiography
Study gas exchange in PACU | up to 24 hours
  SpO2/FiO2
Study gas exchange on day 1 after surgery | on the 1st day after surgery
  SpO2/FiO2
Study gas exchange on day 2 after surgery | on the 2nd day after surgery
  SpO2/FiO2
incidence of postoperative respiratory complications in the month following ENT cancer surgery (eg number of participants with a postoperative respiratory complication) | up to 31 days
  number of participants who had a postoperative respiratory complication within 30 days of surgery: atelectasis, pulmonary oedema, consolidation, pneumothorax, pleural effusion, bronchospasm, pneumonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goel N, Sen IM, Bakshi J. Lung ultrasonography as a tool to guide perioperative atelectasis treatment bundle in head and neck cancer patients undergoing free flap reconstructive surgeries: a preliminary observational study. Braz J Otorhinolaryngol. 2022 Mar-Apr;88(2):204-211. doi: 10.1016/j.bjorl.2020.05.030. Epub 2020 Jul 29. PMID 32800584
- [Background] Touw HR, Parlevliet KL, Beerepoot M, Schober P, Vonk A, Twisk JW, Elbers PW, Boer C, Tuinman PR. Lung ultrasound compared with chest X-ray in diagnosing postoperative pulmonary complications following cardiothoracic surgery: a prospective observational study. Anaesthesia. 2018 Aug;73(8):946-954. doi: 10.1111/anae.14243. Epub 2018 Mar 12. PMID 29529332
- [Background] Zieleskiewicz L, Papinko M, Lopez A, Baldovini A, Fiocchi D, Meresse Z, Boussuges A, Thomas PA, Berdah S, Creagh-Brown B, Bouhemad B, Futier E, Resseguier N, Antonini F, Duclos G, Leone M. Lung Ultrasound Findings in the Postanesthesia Care Unit Are Associated With Outcome After Major Surgery: A Prospective Observational Study in a High-Risk Cohort. Anesth Analg. 2021 Jan;132(1):172-181. doi: 10.1213/ANE.0000000000004755. PMID 32224722
- [Background] Monastesse A, Girard F, Massicotte N, Chartrand-Lefebvre C, Girard M. Lung Ultrasonography for the Assessment of Perioperative Atelectasis: A Pilot Feasibility Study. Anesth Analg. 2017 Feb;124(2):494-504. doi: 10.1213/ANE.0000000000001603. PMID 27669555